CLINICAL TRIAL: NCT03824236
Title: Efficacy, Immunogenicity and Safety Study Evaluating a Fractional (Fx) Booster Dose of GSK Biologicals' Candidate Malaria Vaccine (SB257049) in a Sporozoite Challenge Model in Healthy Malaria-naïve Adults
Brief Title: A Study to Evaluate the Efficacy, Immunogenicity and Safety in a Sporozoite Challenge Model of a Fractional Booster Dose of GSK Biologicals' Candidate Malaria Vaccine Administered to Previously Vaccinated Healthy Malaria-naïve Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: PATH (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 209003; 17337 (Other: IND number)
Record Dates: First submitted 2019-01-29; First posted 2019-01-31 (Actual); Results first posted 2020-05-15 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Malaria
Keywords: Malaria; RTS,S/AS01E vaccine; Fractional dose; Sporozoite challenge
MeSH Terms: conditions — Malaria | interventions — RTS malaria vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- P-Fx group (Experimental): Healthy subjects, between and including 18 and 55 years of age, vaccinated with RTS,S/AS01 vaccine (different doses/formulations) and protected following the first challenge at the time of the MALARIA-092 study (NCT03162614), who received, in the current study, a fractional (Fx) booster dose of RTS,S/AS01E 12 months after completion of the vaccination course in the Malaria-092 study, and underwent sporozoite challenge.
  Interventions: Biological: RTS,S/AS01E (SB257049)
- NP-Fx group (Experimental): Healthy subjects, between and including 18 and 55 years of age, vaccinated with RTS,S/AS01 vaccine (different doses/formulations) and not protected following the first challenge at the time of the MALARIA-092 study (NCT03162614), who received, in the current study, a fractional (Fx) booster dose of RTS,S/AS01E 12 months after completion of the vaccination course in the Malaria-092 study, and underwent sporozoite challenge.
  Interventions: Biological: RTS,S/AS01E (SB257049)
- InfectivityCtrl group (No Intervention): Healthy subjects, between and including 18 and 55 years of age, who did not receive, in the current study, any immunization but underwent sporozoite challenge.

INTERVENTIONS:
Biological: RTS,S/AS01E (SB257049) — Subjects from the P-Fx and NP-Fx groups will receive one Fx booster dose of RTS,S/AS01E at Day 1.
  Arms: NP-Fx group; P-Fx group

SUMMARY:
MALARIA-092 (NCT03162614) study was designed to evaluate the efficacy, immunogenicity and safety of various dose schedules and formulations of GSK Biologicals' candidate malaria vaccine (RTS,S/AS01E) in healthy malaria-naïve subjects aged 18-55 years.

The purpose of this study (follow-up to MALARIA-092 [NCT03162614] study) is to evaluate if protection can be extended with an additional Fx booster dose and if unprotected subjects can be protected following a Fx booster dose.

In this booster study, subjects from MALARIA-092 (NCT03162614) study who completed vaccination and challenge will receive a Fx booster dose of RTS,S/AS01E and undergo a second controlled human malaria infection (CHMI) three to four weeks after vaccination. Additionally, subjects will be newly enrolled and will only undergo the sporozoite challenge as infectivity controls.

ELIGIBILITY:
Inclusion Criteria:

Only for subjects from MALARIA-092 study (NCT03162614):

• Subjects vaccinated and having undergone sporozoite challenge during the primary study (MALARIA-092 [NCT03162614]).

For all subjects:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Written informed consent obtained from the subject prior to performing any study-specific procedure.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Available to participate for the duration of the study.
* Female subjects of non-childbearing potential may be enrolled in the study.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * Has practiced adequate contraception for 30 days prior to Day 1, and has agreed to continue adequate contraception during the entire treatment period and for two months after malaria challenge (only for subjects from the MALARIA-092 study [NCT03162614]).
  * Has practiced adequate contraception for 30 days prior to malaria challenge, and has agreed to continue adequate contraception up to two months after malaria challenge (only for the infectivity control subjects).
  * Has a negative pregnancy test at enrollment.

For the infectivity control subjects:

• Male or female subjects between, and including, 18 and 55 years of age.

Exclusion Criteria:

For all subjects except the infectivity control subjects:

* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine.
* History of anaphylaxis post-vaccination.

For all subjects:

* Use of any investigational or non-registered product other than the study vaccine during the period starting 30 days before Day 1 (Day -29 to Day 1) (for P-Fx and NP-Fx groups)/before the malaria challenge (for infectivity control subjects), or planned use during the study period.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting six months prior to Day 1 (for P-Fx and NP-Fx groups) or malaria challenge (for infectivity control subjects). For corticosteroids, this will mean prednisone ≥20 mg/day, or equivalent. Inhaled and topical steroids are allowed.
* Administration of long-acting immune-modifying drugs at any time during the study period.
* Chronic use of antibiotics with anti-malarial effects.
* Planned administration/administration of a vaccine not foreseen by the study protocol in the period within seven days of Day 1 (for P-Fx and NP-Fx groups) or the malaria challenge (for infectivity control subjects).
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product.
* Seropositive for Human Immunodeficiency Virus, Hepatitis B surface antigen or Hepatitis C Virus.
* Planned travel to malaria endemic areas during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* History of any reaction or hypersensitivity that would prevent the subject from utilizing all of the following: chloroquine, atovaquone/proguanil, artemether/lumefantrine.
* Current use of medications known to cause drug reactions that would prevent the subject from utilizing any of the following: chloroquine, atovaquone/proguanil, artemether/lumefantrine.
* History of severe reactions to mosquito bites.
* Acute disease and/or fever at the time of enrollment.

  * Fever is defined as temperature ≥37.5°C/99.5°F for oral, axillary or tympanic route.
  * Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Hepatomegaly, right upper quadrant abdominal pain or tenderness.
* Any abnormal baseline laboratory screening tests: ALT, AST, creatinine, hemoglobin, platelet count, total WBC, out of normal range.
* Personal history of auto-immune disease.
* Administration of immunoglobulins and/or any blood products during the period starting three months before Day 1 (for P-Fx and NP-Fx groups)/the malaria challenge (for infectivity control subjects), or planned administration during the study period.
* Pregnant or lactating female.
* Female planning to become pregnant or planning to discontinue contraceptive precautions.
* History of chronic alcohol consumption and/or drug abuse.
* History of blood donation within 56 days preceding enrollment.
* Any other significant finding that in the opinion of the investigator would increase the risk of having an adverse outcome from participating in this study.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.
* Evidence of increased cardiovascular disease risk, "moderate" or "high", according to the National Health And Nutrition Examination Survey I (NHANES I) criteria.

Only for infectivity control subjects:

* Previous vaccination against malaria.
* History of splenectomy.
* Family history of congenital or hereditary immunodeficiency.
* Major congenital defects.
* Serious chronic illness.
* History of any neurological disorders or seizures.
* Diagnosed with malaria within the last 5 years (inclusive).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 61 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline (for GlaxoSmithKline; Human Genome Sciences Inc., a GSK Company; Sirtris, a GSK Company; Stiefel, a GSK Company; ViiV Healthcare)
Locations (1):
- GSK Investigational Site, Silver Spring, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Spreng RL, Seaton KE, Lin L, Hilliard S, Horn GQ, Abraha M, Deal AW, Li K, Carnacchi AJ, Feeney E, Shabbir S, Zhang L, Bekker V, Mudrak SV, Dutta S, Mercer LD, Gregory S, King CR, Wille-Reece U, Jongert E, Kisalu NK, Tomaras GD, Dennison SM. Identification of RTS,S/AS01 vaccine-induced humoral biomarkers predictive of protection against controlled human malaria infection. JCI Insight. 2024 Oct 8;9(19):e178801. doi: 10.1172/jci.insight.178801. PMID 39377226
- [Derived] Moon JE, Greenleaf ME, Regules JA, Debois M, Duncan EH, Sedegah M, Chuang I, Lee CK, Sikaffy AK, Garver LS, Ivinson K, Angov E, Morelle D, Lievens M, Ockenhouse CF, Ngauy V, Ofori-Anyinam O; RTS S Malaria Vaccine Working Group. A phase IIA extension study evaluating the effect of booster vaccination with a fractional dose of RTS,S/AS01E in a controlled human malaria infection challenge. Vaccine. 2021 Oct 15;39(43):6398-6406. doi: 10.1016/j.vaccine.2021.09.024. Epub 2021 Sep 27. PMID 34593270

RESULTS

PARTICIPANT FLOW:
Groups:
- Infectivity Control Group: Healthy subjects, between and including 18 and 55 years of age, who did not receive, in the current study, any immunization but underwent sporozoite challenge.
Period: Overall Study
Arm/Group | P-Fx Group | NP-Fx Group | Infectivity Control Group
Started | 25 | 24 | 12
Completed | 25 | 24 | 11
Not Completed | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | P-Fx Group | NP-Fx Group | Infectivity Control Group | Total
Number analyzed (Participants) | 25 | 24 | 12 | 61
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.7 (10.2) | 35.5 (10.1) | 31.7 (10.8) | 34.8 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 10 | 4 | 24
  Male | 15 | 14 | 8 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  AMERICAN INDIAN OR ALASKA NATIVE | 1 | 1 | 0 | 2
  ASIAN | 2 | 1 | 2 | 5
  BLACK OR AFRICAN AMERICAN | 7 | 11 | 4 | 22
  OTHER, Not specified | 0 | 0 | 1 | 1
  WHITE | 15 | 11 | 5 | 31

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Reporting Plasmodium Falciparum (P. Falciparum) Parasitemia (Defined by a Positive Blood Slide) Following Sporozoite Challenge (in All Study Groups Versus Infectivity Controls)
Description: Occurrence of P. falciparum parasitemia (defined by a positive blood slide) following sporozoite challenge. Post-challenge, parasitemia was determined by microscopy of Giemsa-stained thick blood films (smear). Microscopy was performed on thick smears using a validated standard operation procedure. P. falciparum infection was defined as asexual blood stage P. falciparum parasite density greater than (>) 0 detected by blood slide reading. For the analysis of proportion affected (relative risk), all subjects included in the analysis were considered at risk of infection and no censoring or elimination was applied for subjects not completing the entire protocol-defined post-challenge follow-up (Day 50 - 28 days post challenge).
Time Frame: During the sporozoite challenge dose follow-up period (from Day 22 up to Day 50)
Population: Analysis was performed on Per-Protocol Set which included all subjects fulfilling eligibility criteria, who received or not the Fx dose of study vaccine according to protocol, did not report any underlying medical condition influencing the efficacy response, underwent P. falciparum challenge and had available data concerning outcome measures.
Measure: Count of Participants; unit: Participants
Arm/Group | P-Fx Group | NP-Fx Group | Infectivity Control Group
Number analyzed (Participants) | 25 | 24 | 11
Participants | 12 | 11 | 11
Statistical Analysis 1: Comparison: P-Fx Group vs Infectivity Control Group; Efficacy analysis aimed at comparing P. falciparum parasitemia incidence after sporozoite challenge between P-Fx group and the Infectivity Control group; Test type: Other — Vaccine efficacy rate was calculated as 100*(1-RR) with RR=relative risk of developing the disease for vaccinated people (P-Fx Group) compared to unvaccinated people (Infectivity Control Group); p = 0.003, Fisher Exact; Vaccine efficacy rate = 52, 95% CI 2-sided [28 to 68]
Statistical Analysis 2: Comparison: NP-Fx Group vs Infectivity Control Group; Efficacy analysis aimed at comparing P. falciparum parasitemia incidence after sporozoite challenge between NP-Fx group and the Infectivity Control group; Test type: Other — Vaccine efficacy rate was calculated as 100*(1-RR) with RR=relative risk of developing the disease for vaccinated people (NP-Fx Group) compared to unvaccinated people (Infectivity Control Group); p = 0.002, Fisher Exact; Vaccine efficacy rate = 54, 95% CI 2-sided [29 to 70]

2. Secondary Outcome: Time to Onset of P. Falciparum Parasitemia (Defined by a Positive Blood Slide) Following Sporozoite Challenge
Description: For the analyses of time to onset of parasitemia (Kaplan-Meyer and log-rank), time at risk started on first day of challenge. Time at risk was censored on Day 50 (28 days post challenge), drop-out date, start date of anti-malarial treatment or date meeting an endpoint, whichever occured first. Time-at-risk was calculated as: censor date - date challenge + 1.
Time Frame: During the sporozoite challenge period starting at Day 22 (after the vaccine dose administered at Day 1), up to Day 50
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | P-Fx Group | NP-Fx Group | Infectivity Control Group
Number analyzed (Participants) | 12 | 11 | 11
Days | 14.6 (1.9) | 14.1 (1.6) | 11.6 (0.9)

3. Secondary Outcome: Anti- Circumsporozoite (CS) Repeat Region Antibody Concentrations
Description: Anti-CS antibody concentrations are presented as Geometric Mean Concentrations (GMCs), expressed in Enzyme-linked immunosorbent assay Unit per milliliter (EU/mL). The cut-off for the assay was equal to 1.9 EU/mL. GMC calculations are performed by taking the inverse logarithm of the mean of the log concentration transformations. Antibody concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMC calculation.
Time Frame: At Day 1, prior to challenge (Day 22), 28 days post-challenge (Day 50) and at study end (Day 190)
Population: Analysis was performed on Per-Protocol Set which included all subjects fulfilling eligibility criteria, who received the Fx dose according to protocol, underwent P. falciparum challenge and had available immunogenicity data concerning outcome measures. Analysis was not performed on the Infectivity Control Group (no Fx dose being administered).
Measure: Geometric Mean (95% Confidence Interval); unit: EU/mL
Arm/Group | P-Fx Group | NP-Fx Group
Number analyzed (Participants) | 25 | 24
EU/mL
  Day 1: number analyzed (Participants) | 25 | 19
  Day 1 | 32.8 [24.5 to 44.1] | 7.2 [3.9 to 13.4]
  Day 22 | 87.3 [67.0 to 113.9] | 37.3 [23.4 to 59.5]
  Day 50 | 77.8 [59.5 to 101.8] | 25.7 [15.3 to 43.2]
  Day 190: number analyzed (Participants) | 25 | 21
  Day 190 | 49.7 [37.7 to 65.7] | 12.7 [6.9 to 23.4]

4. Secondary Outcome: Anti-Hepatitis B (HBs) Immunoglobulin G (IgG) Antibody Concentrations
Description: Anti-HBs IgG antibody concentrations are presented as Geometric Mean Concentrations (GMCs), expressed in milli-International Unit per milliliter (mIU/mL). The cut-off for the assay was equal to 6.2 mIU/mL. GMC calculations are performed by taking the inverse logarithm of the mean of the log concentration transformations. Antibody concentrations below the cut-off of the assay will be given an arbitrary value of half the cut-off of the assay for the purpose of GMC calculation.
Time Frame: At Day 1, prior to challenge (Day 22), 28 days post-challenge (Day 50) and at study end (Day 190)
Population: as for outcome 3
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | P-Fx Group | NP-Fx Group
Number analyzed (Participants) | 25 | 24
mIU/mL
  Day 1 | 7788 [4822.8 to 12576.4] | 6608.1 [3147.2 to 13874.8]
  Day 22: number analyzed (Participants) | 23 | 24
  Day 22 | 25344.5 [16377.3 to 39221.5] | 29271.3 [18417.1 to 46522.4]
  Day 50 | 21203.1 [14058.2 to 31979.2] | 19894.8 [11569.4 to 34211.1]
  Day 190: number analyzed (Participants) | 24 | 22
  Day 190 | 11593.9 [7446.0 to 18052.6] | 9092.5 [4652.8 to 17768.4]

5. Secondary Outcome: Number of Subjects With Any Solicited Local Adverse Events (AEs) in the Booster Vaccination Groups
Description: Solicited local AEs assessed are erythema, pain and swelling. Any occurrence of AE regardless of intensity grade are reported. Any Erythema or any Swelling symptom = any symptom recorded with a surface diameter greater than 0 millimeter.
Time Frame: Within 7 days after vaccination (day of vaccination and 6 subsequent days) in the booster vaccination groups
Population: Analysis was performed on Intent-To-Treat Set, which included all subjects from the P-Fx and NP-Fx groups who received the Fx dose of the study vaccine and with the symptoms sheet documented.
Measure: Count of Participants; unit: Participants
Arm/Group | P-Fx Group | NP-Fx Group
Number analyzed (Participants) | 25 | 24
Participants
  Erythema | 8 | 4
  Pain | 11 | 10
  Swelling | 4 | 4

6. Secondary Outcome: Number of Subjects With Any Solicited General AEs in the Booster Vaccination Groups
Description: Solicited general AEs assessed are fatigue, gastrointestinal symptoms (nausea, vomiting, diarrhea and/or abdominal pain), headache and fever. Any occurrence of symptom regardless of intensity grade and relationship to the vaccination. Fever was defined as temperature equal or greater than 37.5 °C (preferably oral route measure).
Time Frame: Within 7 days after vaccination (day of vaccination and 6 subsequent days) in the booster vaccination groups
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | P-Fx Group | NP-Fx Group
Number analyzed (Participants) | 25 | 24
Participants
  Fatigue | 7 | 4
  Gastrointestinal symptoms | 2 | 0
  Headache | 6 | 5
  Fever | 3 | 0

7. Secondary Outcome: Number of Subjects With Any Unsolicited AEs After Vaccination, in the Booster Vaccination Groups
Description: An unsolicited adverse event is any untoward medical occurrence in a clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. An unsolicited adverse event is any event reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Up to 21 days after booster vaccination period (day of vaccination and 20 subsequent days), after booster vaccination
Population: Analysis was performed on Intent-To-Treat Set, which included all subjects from the P-Fx and NP-Fx groups who received the Fx dose of the study vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | P-Fx Group | NP-Fx Group
Number analyzed (Participants) | 25 | 24
Participants | 5 | 1

8. Secondary Outcome: Number of Subjects With Any Unsolicited AEs After Challenge, in All Study Groups
Description: An adverse event is any untoward medical occurrence in a clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Within 29 days after challenge (day of challenge and 28 subsequent days)
Population: Analysis was performed on Intent-To-Treat Set, which included all subjects who received at least one dose of study vaccine. All challenged infectivity controls were also included in this analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | P-Fx Group | NP-Fx Group | Infectivity Control Group
Number analyzed (Participants) | 25 | 24 | 12
Participants | 19 | 19 | 12

9. Secondary Outcome: Number of Subjects With AEs of Specific Interest (Potential Immune-mediated Diseases [pIMDs] and Meningitis), in All Study Groups
Description: AEs of specific interest are potential immune-mediated diseases (pIMDs) and meningitis. pIMDs are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune etiology.
Time Frame: From Day 1 up to study conclusion (Day 190)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | P-Fx Group | NP-Fx Group | Infectivity Control Group
Number analyzed (Participants) | 25 | 24 | 12
Participants | 0 | 0 | 0

10. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) (Any, Fatal or Related to Investigational Vaccine) During the Whole Study Period, in All Study Groups
Description: An SAE is any untoward medical occurrence that results in death, is life threatening, requires hospitalization or prolongation of hospitalization, results in disability/incapacity or is a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: From Day 1 up to study conclusion (Day 190)
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | P-Fx Group | NP-Fx Group | Infectivity Control Group
Number analyzed (Participants) | 25 | 24 | 12
Participants
  Any SAEs | 2 | 0 | 0
  Related SAEs | 0 | 0 | 0
  Fatal SAEs | 0 | 0 | 0

11. Secondary Outcome: Number of Subjects With Abnormal Laboratory Values
Description: Biochemistry (Alanine Aminotransferase [ALT], Aspartate Aminotransferase [AST] and Creatinine) and hematological (Hemoglobin, Platelets, White Blood Cells [WBC] decrease and WBC increase) laboratory values were presented according to toxicity grading scales and tabulated by group. Grading scale adapted from FDA guidance for industry: toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventive vaccine clinical trials (September 2007).
Time Frame: At screening, Day(D)1, D8, D22 (day of first parasitemia) and D50 (28 days post-challenge) for the booster vaccination groups; and at screening, D22 (day of first parasitemia) and D50 (28 days post-challenge) for the infectivity control subjects
Population: as for outcome 8
Measure: Count of Participants; unit: Participants
Arm/Group | P-Fx Group | NP-Fx Group | Infectivity Control Group
Number analyzed (Participants) | 25 | 24 | 12
Participants
  ALT, Screening, Grade 0 | 24 | 23 | 11
  ALT, Screening, Grade 1 | 1 | 1 | 1
  ALT, Day 1, Grade 0: number analyzed (Participants) | 25 | 24 | 0
  ALT, Day 1, Grade 0 | 25 | 23 |
  ALT, Day 1, Grade 1: number analyzed (Participants) | 25 | 24 | 0
  ALT, Day 1, Grade 1 | 0 | 1 |
  ALT, Day 8, Grade 0: number analyzed (Participants) | 25 | 24 | 0
  ALT, Day 8, Grade 0 | 24 | 24 |
  ALT, Day 8, Grade 1: number analyzed (Participants) | 25 | 24 | 0
  ALT, Day 8, Grade 1 | 1 | 0 |
  ALT, Day 22, Grade 0 | 23 | 23 | 12
  ALT, Day 22, Grade 1 | 2 | 1 | 0
  ALT, Day 50, Grade 0: number analyzed (Participants) | 25 | 24 | 11
  ALT, Day 50, Grade 0 | 23 | 22 | 10
  ALT, Day 50, Grade 1: number analyzed (Participants) | 25 | 24 | 11
  ALT, Day 50, Grade 1 | 2 | 2 | 1
  AST, Screening, Grade 0 | 25 | 24 | 11
  AST, Screening, Grade 1 | 0 | 0 | 1
  AST, Day 1, Grade 0: number analyzed (Participants) | 25 | 24 | 0
  AST, Day 1, Grade 0 | 24 | 24 |
  AST, Day 1, Grade 1: number analyzed (Participants) | 25 | 24 | 0
  AST, Day 1, Grade 1 | 1 | 0 |
  AST, Day 8, Grade 0: number analyzed (Participants) | 25 | 24 | 0
  AST, Day 8, Grade 0 | 24 | 24 |
  AST, Day 8, Grade 1: number analyzed (Participants) | 25 | 24 | 0
  AST, Day 8, Grade 1 | 1 | 0 |
  AST, Day 22, Grade 0 | 25 | 23 | 12
  AST, Day 22, Grade 1 | 0 | 1 | 0
  AST, Day 50, Grade 0: number analyzed (Participants) | 25 | 24 | 11
  AST, Day 50, Grade 0 | 25 | 24 | 10
  AST, Day 50, Grade 1: number analyzed (Participants) | 25 | 24 | 11
  AST, Day 50, Grade 1 | 0 | 0 | 1
  Creatinine, Screening, Grade 0 | 25 | 24 | 12
  Creatinine, Day 1, Grade 0: number analyzed (Participants) | 25 | 24 | 0
  Creatinine, Day 1, Grade 0 | 25 | 24 |
  Creatinine, Day 8, Grade 0: number analyzed (Participants) | 25 | 24 | 0
  Creatinine, Day 8, Grade 0 | 25 | 24 |
  Creatinine, Day 22, Grade 0 | 25 | 24 | 12
  Creatinine, Day 50, Grade 0: number analyzed (Participants) | 25 | 24 | 11
  Creatinine, Day 50, Grade 0 | 25 | 24 | 11
  Hemoglobin, Screening, Grade 0 | 24 | 23 | 12
  Hemoglobin, Screening, Grade 1 | 1 | 1 | 0
  Hemoglobin, Day 1, Grade 0: number analyzed (Participants) | 25 | 24 | 0
  Hemoglobin, Day 1, Grade 0 | 25 | 22 |
  Hemoglobin, Day 1, Grade 1: number analyzed (Participants) | 25 | 24 | 0
  Hemoglobin, Day 1, Grade 1 | 0 | 2 |
  Hemoglobin, Day 8, Grade 0: number analyzed (Participants) | 25 | 24 | 0
  Hemoglobin, Day 8, Grade 0 | 25 | 22 |
  Hemoglobin, Day 8, Grade 1: number analyzed (Participants) | 25 | 24 | 0
  Hemoglobin, Day 8, Grade 1 | 0 | 2 |
  Hemoglobin, Day 22, Grade 0 | 23 | 21 | 10
  Hemoglobin, Day 22, Grade 1 | 2 | 2 | 2
  Hemoglobin, Day 22, Grade 2 | 0 | 1 | 0
  Hemoglobin, Day 50, Grade 0: number analyzed (Participants) | 25 | 24 | 11
  Hemoglobin, Day 50, Grade 0 | 23 | 22 | 10
  Hemoglobin, Day 50, Grade 1: number analyzed (Participants) | 25 | 24 | 11
  Hemoglobin, Day 50, Grade 1 | 2 | 2 | 1
  Platelets, Screening, Grade 0 | 24 | 24 | 12
  Platelets, Screening, Grade 1 | 1 | 0 | 0
  Platelets, Day 1, Grade 0: number analyzed (Participants) | 25 | 24 | 0
  Platelets, Day 1, Grade 0 | 24 | 24 |
  Platelets, Day 1, Grade 2: number analyzed (Participants) | 25 | 24 | 0
  Platelets, Day 1, Grade 2 | 1 | 0 |
  Platelets, Day 8, Grade 0: number analyzed (Participants) | 25 | 24 | 0
  Platelets, Day 8, Grade 0 | 25 | 24 |
  Platelets, Day 22, Grade 0 | 24 | 24 | 12
  Platelets, Day 22, Grade 1 | 1 | 0 | 0
  Platelets, Day 50, Grade 0: number analyzed (Participants) | 25 | 24 | 11
  Platelets, Day 50, Grade 0 | 25 | 24 | 11
  WBC Decrease, Screening, Grade 0 | 24 | 24 | 12
  WBC Decrease, Screening, Grade 1 | 1 | 0 | 0
  WBC Decrease, Day 1, Grade 0: number analyzed (Participants) | 25 | 24 | 0
  WBC Decrease, Day 1, Grade 0 | 24 | 22 |
  WBC Decrease, Day 1, Grade 1: number analyzed (Participants) | 25 | 24 | 0
  WBC Decrease, Day 1, Grade 1 | 0 | 2 |
  WBC Decrease, Day 1, Grade 2: number analyzed (Participants) | 25 | 24 | 0
  WBC Decrease, Day 1, Grade 2 | 1 | 0 |
  WBC Decrease, Day 8, Grade 0: number analyzed (Participants) | 25 | 24 | 0
  WBC Decrease, Day 8, Grade 0 | 25 | 23 |
  WBC Decrease, Day 8, Grade 1: number analyzed (Participants) | 25 | 24 | 0
  WBC Decrease, Day 8, Grade 1 | 0 | 1 |
  WBC Decrease, Day 22, Grade 0 | 25 | 24 | 12
  WBC Decrease, Day 50, Grade 0: number analyzed (Participants) | 25 | 24 | 11
  WBC Decrease, Day 50, Grade 0 | 24 | 23 | 11
  WBC Decrease, Day 50, Grade 1: number analyzed (Participants) | 25 | 24 | 11
  WBC Decrease, Day 50, Grade 1 | 1 | 1 | 0
  WBC Increase, Screening, Grade 0 | 25 | 24 | 12
  WBC Increase, Day 1, Grade 0: number analyzed (Participants) | 25 | 24 | 0
  WBC Increase, Day 1, Grade 0 | 25 | 24 |
  WBC Increase, Day 8, Grade 0: number analyzed (Participants) | 25 | 24 | 0
  WBC Increase, Day 8, Grade 0 | 25 | 24 |
  WBC Increase, Day 22, Grade 0 | 25 | 24 | 12
  WBC Increase, Day 50, Grade 0: number analyzed (Participants) | 25 | 24 | 11
  WBC Increase, Day 50, Grade 0 | 25 | 24 | 11

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected within the 7-day post-booster period. Unsolicited AEs were collected within the 21-day post-booster or within the 29-day post-challenge period. SAEs were collected from Day 1 up to study conclusion (Day 190).
Arm/Group | P-Fx Group | NP-Fx Group | Infectivity Control Group
All-Cause Mortality (participants affected / at risk) | 0/25 | 0/24 | 0/12
Serious Adverse Events (participants affected / at risk) | 2/25 | 0/24 | 0/12
Other Adverse Events (participants affected / at risk) | 21/25 | 22/24 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P-Fx Group (N=25) | NP-Fx Group (N=24) | Infectivity Control Group (N=12)
Hypobarism (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — The same subject reported both injury and road traffic accident.
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) — The same subject reported both injury and road traffic accident.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | P-Fx Group (N=25) | NP-Fx Group (N=24) | Infectivity Control Group (N=12)
Injection site pain (General disorders) | 11 (11) | 10 (10) | 0 (0)
Fatigue (General disorders) | 11 (11) | 7 (7) | 1 (1)
Injection site erythema (General disorders) | 8 (8) | 4 (4) | 0 (0)
Injection site swelling (General disorders) | 4 (4) | 4 (4) | 0 (0)
Chills (General disorders) | 3 (4) | 2 (2) | 0 (0)
Feeling hot (General disorders) | 2 (2) | 2 (2) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 1 (1) | 0 (0)
Malaise (General disorders) | 1 (1) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 1 (1) | 0 (0)
Thirst (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 12 (12) | 11 (11) | 11 (11)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 5 (5) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Muscle tightness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Joint warmth (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 9 (11) | 8 (8) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 3 (3) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Gastrointestinal disorder (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (4) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-09-26): https://cdn.clinicaltrials.gov/large-docs/36/NCT03824236/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-20): https://cdn.clinicaltrials.gov/large-docs/36/NCT03824236/SAP_001.pdf